CLINICAL TRIAL: NCT02249793
Title: Exploratory Study in Healthy Volunteers to Define Circadian Relationships Between Social Behavior, Blood Pressure and Metabolomics
Brief Title: Exploratory Study of Circadian Relationships Between Social Behavior, Blood Pressure and Metabolomics
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Ginger.io (Industry)
Responsible Party: Principal Investigator, Carsten Skarke, MD, Research Assistant Professor, University of Pennsylvania
Other Study IDs: 817759
Record Dates: First submitted 2014-03-25; First posted 2014-09-26 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Healthy
Keywords: circadian; oscillation; clock; human; social behavior; cell phone with internet access (so-called smartphone); social sensing; behavioral feature; Ginger.io; blood pressure; metabolism; metabolomics; gut bacteria; microbiome
MeSH Terms: conditions — Social Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, urine, stool, and mucosal swabs from nose, mouth and rectum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Healthy volunteers

SUMMARY:
As citizens of the information age, humans leave digital traces of behavior in their communication and movement patterns through our cell phone. The Global Positioning System (GPS) technology tracks the way persons commute to school or work or when visiting family and friends. Circadian rhythmicity describes the concept that many of the bodily functions follow a roughly 24-hour rhythm. Usually, the ability to do concentrated and focused work is best during daytime while humans rest and sleep during nighttime. The current study wishes to look for a relationship between patterns in participants' cell phone use (Android only at this point) and several of their bodily functions.

DETAILED DESCRIPTION:
Cell phones with internet access (so-called smartphones) represent a rich source for user activity data. Each time one places a call, sends a text message, or uses an app, a data trace is being produced which overall reflects the user's social activity and behavior. This data is called 'social sensing data'. Researchers connected this type of data to the health status of the person operating the cell phone. An example is that an outbreak of seasonal flu may lead to fewer calls and text messages among cell phone users. Thus, the social sensing data may show for example how severe an outbreak is and how fast it is spreading.

"Circadian rhythmicity" describes the concept that many of the bodily functions follow a roughly 24-hour rhythm. Usually, the ability to do concentrated and focused work is best during daytime while rest and sleep occurs during nighttime. A disturbance of this pattern, for example by regular nightshift work, may lead to an increased disease risk, such as for the cardiovascular system, the heart and blood vessels. Natural factors within a body produce our 24-hour rhythm. This rhythm is affected by outside cues such as sunlight. Jet lag is a short-term form of a disturbed 24-hour rhythm. When a person travels fast through several time zones, by plane for example from the East to the West Coast of the US, s/he arrives with a time difference of 3 hours. Upon arrival, the body runs still at East Coast time, but is exposed to the environmental cues following the West Coast time, which may make the person feel groggy and disoriented at first. Within a couple of days the body time usually adjusts and the complaints discontinue.

The current study wishes to look for a relationship between patterns in the participant's cell phone use (Android only at this point) and several of the bodily functions. As bodily functions the investigators will measure blood pressure and breakdown products (metabolites) in urine, blood and saliva samples. The investigators will collect stool samples and use swabs to collect the microbes inhabiting the mouth as well as the rectum. The investigators will also measure messenger ribonucleic acid (mRNA), messenger products of the participant's heritable information, in the blood. A cell phone application called "Ginger.io" will collect the participants' cell phone usage information. This application will also ask the participant several questions during the installation, during participation as well as at the end. Furthermore, the investigators will ask the participant about the dietary intake and habits.

The aim is to learn how the 24-hour rhythm is connected to the social activity and behavior as well as blood pressure and metabolites as markers for the health status.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must be in good health as based on medical history, physical examination, vital signs, and laboratory tests as deemed by PI;
* Volunteers are capable of giving informed consent;
* 25-35 years of age;
* Own a cell phone with internet access (smartphone with Android operating system only at this point) which installs the social sensing application ginger.io;
* Non-smoking;
* Male subjects only if feasible during recruitment; and
* In case female volunteers are invited to enroll: non-pregnant, female subjects must consent to a urine pregnancy test.

Exclusion Criteria:

* Recent travel across time zones (within the past month);
* Planned travel across time zones during the planned study activities;
* Volunteers with irregular work hours, e.g. night shifts.
* Use of illicit drugs;
* Subjects, who have received an experimental drug, used an experimental medical device within 30 days prior to screening, or who gave a blood donation of ≥ one pint within 8 weeks prior to screening.
* Subjects with any abnormal laboratory value or physical finding that according to the investigator may interfere with interpretation of the study results, be indicative of an underlying disease state, or compromise the safety of a potential subject.

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2014-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Skarke, MD, Principal Investigator — University of Pennsylvania; Garret A FitzGerald, MD, Principal Investigator — University of Pennsylvania; Aalim Weljie, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Institute for Translational Medicine and Therapeutics (ITMAT), University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Skarke C, Lahens NF, Rhoades SD, Campbell A, Bittinger K, Bailey A, Hoffmann C, Olson RS, Chen L, Yang G, Price TS, Moore JH, Bushman FD, Greene CS, Grant GR, Weljie AM, FitzGerald GA. A Pilot Characterization of the Human Chronobiome. Sci Rep. 2017 Dec 7;7(1):17141. doi: 10.1038/s41598-017-17362-6. PMID 29215023
- See also: Zenodo data repository — https://zenodo.org/communities/human-chronobiome/?page=1&size=20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Started 9/24/14, Ended 3/11/15 located at the Clinical and Translational Research Center, CTRC located at the University of Pennsylvania Hospital
Groups:
- Session 1, 48-hour: Healthy volunteers; The observation time for the biosensor-derived data was a total of four months with two 48-hour sessions (Session 1 & 2) scheduled two weeks apart to extend the biosensor platform by ambulatory blood pressure monitoring (ABPM) and timestamped dietary intake (SmartIntake) as well as by collection of timed biospecimens for multiomics analysis at 12-hour intervals.
Period: Session 1, 48-hours Healthy Volunteers
Arm/Group | Session 1, 48-hour
Started | 6
Completed | 6
Not Completed | 0
Period: Session 2, 48-Hours Healthy Volunteers
Arm/Group | Session 1, 48-hour
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Male Healthy Volunteers: Males
Arm/Group | Male Healthy Volunteers
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Calls and Text Messages
Description: Aggregate communication as behavioral features has been collected using the cell phone data streams.
Time Frame: 3-4 months
Measure: Mean (Full Range); unit: Calls and text messages
Arm/Group | Study Group
Number analyzed (Participants) | 6
Calls and text messages
  Awake | 18.7 [0 to 166]
  Sleeping | 0.9 [0 to 84]

2. Primary Outcome: Changes Over Time in Ambulatory Blood Pressure - Systolic Blood Pressure
Description: Ambulatory blood pressure monitoring
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Study Group
Number analyzed (Participants) | 6
mmHg
  Difference Day versus Night | 20.7 (3.9)
  Awake | 126.1 (10.6)
  Asleep | 106.8 (11.6)

3. Primary Outcome: Percentage of Total Metabolites
Description: Percentage of metabolites displaying different abundances in biosamples collected during the morning hours versus evening hours. Analysis was performed for all participants as a group.
Time Frame: 48 hours
Measure: Number; unit: percent
Arm/Group | Study Group
Number analyzed (Participants) | 6
percent
  Plasma metabolome | 5.4
  Saliva metabolome | 5.6

4. Primary Outcome: Mobility Radius
Description: The approximate radius of an imaginary circle encompassing the various locations that a user has traveled across on a particular day (in miles)
Time Frame: 3-4 months
Measure: Mean (Full Range); unit: miles
Arm/Group | Study Group
Number analyzed (Participants) | 6
miles | 6.8 [0 to 193.4]

5. Primary Outcome: Calls
Description: Number of phone calls placed and received
Time Frame: 3-4 months
Measure: Mean (Full Range); unit: Calls
Arm/Group | Study Group
Number analyzed (Participants) | 6
Calls
  Awake | 2.7 [0 to 48]
  Sleeping | 0.1 [0 to 10]

6. Primary Outcome: Changes Over Time in Ambulatory Blood Pressure - Diastolic Blood Pressure
Description: Ambulatory blood pressure monitoring
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Study Group
Number analyzed (Participants) | 6
mmHg
  Difference Day versus Night | 20.7 (3.3)
  Awake | 78.5 (9.1)
  Asleep | 58.8 (10.2)

7. Primary Outcome: Unanswered Calls
Description: The number of calls unanswered.
Time Frame: 3-4 months
Measure: Mean (Full Range); unit: Unanswered calls
Arm/Group | Study Group
Number analyzed (Participants) | 6
Unanswered calls
  Awake | 0.6 [0 to 9]
  Sleeping | 0.03 [0 to 2]

8. Primary Outcome: Unique Contacts
Description: The total number of unique individuals with whom a participant interacted through phone calls or sms messages indicating interaction diversity
Time Frame: 3-4 months
Measure: Mean (Full Range); unit: Unique contacts
Arm/Group | Study Group
Number analyzed (Participants) | 6
Unique contacts
  Awake | 7.2 [0 to 71]
  Sleeping | 0.5 [0 to 29]

9. Primary Outcome: Call Duration
Description: The duration of calls (made + received)
Time Frame: 3-4 months
Measure: Mean (Full Range); unit: Seconds
Arm/Group | Study Group
Number analyzed (Participants) | 6
Seconds
  Awake | 820.4 [0 to 16590]
  Sleeping | 22.0 [0 to 3162]

10. Primary Outcome: Text Message Length
Description: The total length of all sms messages (sent + received) in characters
Time Frame: 3-4 months
Measure: Mean (Full Range); unit: n (characters)
Arm/Group | Study Group
Number analyzed (Participants) | 6
n (characters)
  Awake | 868.0 [0 to 14840]
  Sleeping | 47.0 [0 to 3089]

11. Primary Outcome: Text Messages
Description: The number of sms messages (sent + received)
Time Frame: 3-4 months
Measure: Mean (Full Range); unit: messages
Arm/Group | Study Group
Number analyzed (Participants) | 6
messages
  Awake | 16.0 [0 to 166]
  Sleeping | 0.8 [0 to 75]

12. Secondary Outcome: Self-reported Sleep Times [Survey]
Description: Cell phone administered survey where participants indicated start and end of sleep times. From this the total hours of sleep per night was calculated.
Time Frame: 3-4 months
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Session 1, 48-hour
Number analyzed (Participants) | 6
hour | 7.6 (2.9)

13. Secondary Outcome: Time Asleep
Description: Hours asleep per each 24 hour period measured by actigraphy
Time Frame: 3-4 months
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Study Group
Number analyzed (Participants) | 6
hours | 7.931449224 (0.7044404472)

14. Secondary Outcome: Physical Activity
Description: Difference in locomotion between wake and sleep times
Time Frame: 3-4 months
Measure: Mean (Full Range); unit: Counts/min
Arm/Group | Study Group
Number analyzed (Participants) | 6
Counts/min
  Awake | 1904.0 [0 to 55757.7]
  Sleeping | 307.2 [0 to 29642.7]

15. Secondary Outcome: Changes Over Time in Nutrient Intake - Energy
Description: Nutrient intake will be measured using food photography
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: Kcals
Arm/Group | Study Group
Number analyzed (Participants) | 6
Kcals
  Session 1 | 1967 (488)
  Session 2 | 1609 (601)

16. Secondary Outcome: Changes Over Time in Ribonucleic Acids (RNA) - ARNTL (BMAL1) Normalized to GAPDH
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: relative expression
Arm/Group | Study Group
Number analyzed (Participants) | 6
relative expression
  Morning | 23.3 (13.5)
  Evening | 17.9 (9.4)

17. Secondary Outcome: Genera Displaying Different Abundances Measured During Morning Versus Evening Hours in the Oral Microbiome
Description: Analysis was performed for all participants as a group.
Time Frame: 48 hours
Measure: Number; unit: genera
Arm/Group | Study Group
Number analyzed (Participants) | 6
genera | 3

18. Secondary Outcome: Proteins Displaying Different Abundances Measured in the Morning Versus Evening Hours
Description: Analysis was performed for all participants as a group.
Time Frame: 48 hours
Measure: Number; unit: Proteins
Arm/Group | Study Group
Number analyzed (Participants) | 6
Proteins | 2

19. Secondary Outcome: Changes Over Time in Kidney Function
Time Frame: 48 hours
Population: Kidney function was done to evaluate healthy volunteers during Session 1 and 2. Delta was calculated between Session 1 and 2 and averaged across subjects. Note that values for session1 was missing for two subjects, meaning that below reported mean and standard deviation reflect changes for four subjects.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Session 1, 48-hour
Number analyzed (Participants) | 6
mg/dL | 12.925 (115.468246)

ADVERSE EVENTS:
Time Frame: 1 year
Description: All non serious AE were resolved, Serious AE: None
Groups:
- Healthy Volunteers: Males
Arm/Group | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers (N=6)
headache (General disorders) | 1 (2) — 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2014-07-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT02249793/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2014-07-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT02249793/Prot_SAP_001.pdf